CLINICAL TRIAL: NCT00805649
Title: Combined Therapy in ARMD - Retrospective Case Series
Brief Title: Combined Therapy in Age-Related Macular Degeneration (ARMD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Michael Koss, PI, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-KTAMD-2008
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: ARMD; combined therapy; efficacy; safety
MeSH Terms: conditions — Macular Degeneration | interventions — Dexamethasone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): eyes with predominately classic lesions
  Interventions: Procedure: Low fluorescence Photodynamic therapy; Procedure: core pars plana vitrectomy; Drug: dexamethasone; Drug: bevacizumab
- 2 (Experimental): eyes with occult lesions
  Interventions: Drug: bevacizumab; Procedure: core pars plana vitrectomy; Drug: triamcincolone

INTERVENTIONS:
Procedure: Low fluorescence Photodynamic therapy — 42 J/cm2 for 72 sec
  Arms: 1
Procedure: core pars plana vitrectomy — 24 hours after photodynamic therapy, 1.5 mL core pars plana vitrectomy
  Arms: 1
Drug: dexamethasone — intravitreal injection of 0.8 mg dexamethasone
  Arms: 1
Drug: bevacizumab — intravitreal injection of 1.25 mg bevacizumab
Procedure: core pars plana vitrectomy — 0.4 mL core pars plana vitrectomy
  Arms: 2
Drug: triamcincolone — intravitreal injection of 8 mg triamcincolone
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy of combined intravitreal therapy with or without prior photodynamic therapy in patients with wet age-related macular degeneration (AMD).

In patients with wet AMD, a significant improvement in vision was observed after combined intravitreal therapy with or without prior photodynamic therapy. Both the pharmacological effects of the drugs and the physiological effects of the pars plana vitrectomy (posterior vitreous detachment, liquefaction, and oxygen redistribution) may have contributed to the long-term sustainability of the therapeutic benefits.

DETAILED DESCRIPTION:
This prospective study of a case series included eyes with predominantly classic lesions (Group 1; n = 52) and eyes with occult lesions (Group 2; n = 106). Patients with predominantly classic lesions received low fluorescence photodynamic therapy (42 J/cm2 for 72 sec), followed by, 24 hours later, a 1.5 mL core pars plana vitrectomy with intravitreal injection of dexamethasone (0.8 mg) and bevacizumab (1.25 mg). Patients with occult lesions received a 0.4 mL core pars plana vitrectomy with intravitreal injection of triamcinolone (8 mg) and bevacizumab (1.25 mg). At baseline and follow-up examinations, the best-corrected visual acuity (BCVA; logMar), central macular thickness (optical coherence tomography), intraocular pressure (IOP; Goldmann tonometry) were determined. In addition, the need for retreatment was assessed, and adverse events were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Wet age related macular degeneration

Exclusion Criteria:

* Opacities in lens or cornea
* Ongoing intraocular inflammation
* Trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | at the day of exam
Central macular thickness | at the day of exam

CONTACTS AND LOCATIONS:
Locations (1):
- Abteilung für Netzhaut und Glaskörperchirurgie, Frankfurt am Main, Hesse, Germany